CLINICAL TRIAL: NCT06910956
Title: Deep Learning Using Routine Chest X-Rays and Electronic Medical Record Data to Identify High Risk Patients for Lung Cancer Screening CT
Brief Title: Deep Learning Using Chest X-Rays to Identify High Risk Patients for Lung Cancer Screening CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard Risk Management Foundation (Other)
Responsible Party: Principal Investigator, Michael T. Lu, MD, MPH, Associate Chair, Imaging Science, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2023P002872
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer; Health Screening; Early Cancer Detection; Deep Learning
Keywords: Deep learning; AI; Chest x-ray
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: CXR-LC
- Non-Intervention (No Intervention)

INTERVENTIONS:
Other: CXR-LC — Alert to provider to discuss lung cancer screening CT eligibility, for patients considered at high risk of lung cancer based on CXR-LC AI tool.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to evaluate whether an AI tool that alerts providers to patients at high 6-year risk of lung cancer based on their chest x-ray images will improve lung cancer screening CT participation. The main question it aims to answer is: Does the AI tool improve lung cancer screening CT participation at 6 months after the baseline outpatient visit

The intervention is an alert to the provider to discuss lung cancer screening CT eligibility, for patients considered at high risk of lung cancer based on CXR-LC AI tool.

If there is a comparison group: Researchers will compare intervention and non-intervention arms to determine if lung cancer screen CT participation increases.

ELIGIBILITY:
Major Inclusion Criteria:

* Scheduled outpatient appointment with participating provider.
* 50- to 77-year-old who currently or formerly smoked, to include persons potentially eligible for lung screening based on Medicare guidelines.
* Recent (within 2 years) PA chest radiograph.

Exclusion Criteria:

• History or signs/symptoms of lung cancer. Recent (within 2 years) chest CT. Clinical indication for chest CT beyond lung cancer screening.

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion completing Lung Cancer screening CT in 6 months after visit | 6 months
  To assess impact on lung cancer screening CT participation (defined as completing lung cancer screening CT) in the 6 months after the baseline visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu MT, Raghu VK, Mayrhofer T, Aerts HJWL, Hoffmann U. Deep Learning Using Chest Radiographs to Identify High-Risk Smokers for Lung Cancer Screening Computed Tomography: Development and Validation of a Prediction Model. Ann Intern Med. 2020 Nov 3;173(9):704-713. doi: 10.7326/M20-1868. Epub 2020 Sep 1. PMID 32866413
- [Background] Lee JH, Lee D, Lu MT, Raghu VK, Park CM, Goo JM, Choi SH, Kim H. Deep Learning to Optimize Candidate Selection for Lung Cancer CT Screening: Advancing the 2021 USPSTF Recommendations. Radiology. 2022 Oct;305(1):209-218. doi: 10.1148/radiol.212877. Epub 2022 Jun 14. PMID 35699582
- [Background] Raghu VK, Walia AS, Zinzuwadia AN, Goiffon RJ, Shepard JO, Aerts HJWL, Lennes IT, Lu MT. Validation of a Deep Learning-Based Model to Predict Lung Cancer Risk Using Chest Radiographs and Electronic Medical Record Data. JAMA Netw Open. 2022 Dec 1;5(12):e2248793. doi: 10.1001/jamanetworkopen.2022.48793. PMID 36576736